CLINICAL TRIAL: NCT04652466
Title: Comparison of Fiberoptic Bronchoscopy and Ultrasound Imaging to Validate I-gel Placement in Pediatric Patients
Brief Title: Ultrasound Imaging to Validate I-gel Placement in pediatrıc Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Faruk Cicekci, principal investigator, Selcuk University
Other Study IDs: farukcicekci2
Record Dates: First submitted 2020-11-26; First posted 2020-12-03 (Actual); Last update posted 2020-12-03 (Actual); Status verified 2020-11

CONDITIONS: Ultrasound Imaging; Supraglottic Airway Device; Fiberoptic Bronchoscopy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: farukcicekci2 — To compare the incidence of for I-Gel malposition between USG and FOB, and to find the correlation between I-Gel's USG and FOB-detected malposition

SUMMARY:
For nearly half a century, supraglottic airway devices (SGA) have been used in pediatric patients, which are more practical than face masks, facilitate oxygenation and ventilation without the need for endotracheal intubation, and less invasive than endotracheal tubes. I-Gel is a supraglottic airway management device introduced in 2007, made of a medical grade thermoplastic elastomer, designed to create a non-inflatable, anatomical seal in the pharyngeal, laryngeal and perilaryngeal structures that prevents compression trauma. Recently, the use of I-Gel has become popular in children undergoing surgery that does not require muscle relaxation. It is important to place an I-Gel in the most appropriate position in order to provide adequate ventilation and prevent complications such as mucosal injury, glottic ptosis, and gastric insufflation with potential aspiration. Successful placement is usually clinically assessed by a capnogram with endtidal carbon dioxide (ETCO2) value, visual examination and auscultation with appropriate chest elevation, absence of oropharyngeal leakage at 20 cm H2O peak inspiratory pressure. Although Fiberoptic Bronchoscope (FOB) is accepted as the preferred verification tool for direct visualization, some studies on I-Gel position using FOB reported that I-Gel placement should be repositioned in some children (12.8-49%). Ultrasonography (USG), which has recently entered the practice of upper airway examination, has become a valuable, non-invasive, simple and portable technology for evaluating airway management even in upper airway anatomy impaired by pathology or trauma. The aim of this study is to compare the use of USG with the FOB to evaluate I-Gel placement in pediatric patients. The primary endpoint is to compare the incidence of for I-Gel malposition between USG and FOB. Secondary endpoints are to find the correlation between I-Gel's USG and FOB-detected malposition and to determine the diagnostic performance of the USG.

DETAILED DESCRIPTION:
The population of the study was created from the parents of pediatric patients who were scheduled for elective pediatric surgery under general anesthesia between December 2020 and February 2021 at Selcuk University Department of Anesthesiology and Reanimation. All patients were monitored with standard monitoring (ECG, non-invasive blood pressure, SpO2, ETCO2, Ppeak), after a minimum of 2 minutes of preoxygenation, mask ventilation was performed with 6-7% sevoflurane at the beginning of general anesthesia induction. Intravenous vein access was provided, and according to standard procedures; propofol 3.5 mg.kg 1, fentanyl 1 mg.kg 1 iv and remifentanil 0.1 mcg kg min 1 infusion was administered, but neuromuscular blocker was not used. The choice of the size of the I-Gel was selected according to the manufacturer's recommendations (size 1: 2-5 kg, size 1.5: 5 to 12 kg, size 2: 10 to 25 kg). Adequate anesthesia depth was confirmed by loss of eyelash reflex, symmetrical small pupils and absence of swallowing, and was guided gently along the hard palate by the 1st anesthesiologist until resistance was felt, with the I-Gel opening facing the applicator. If the patient did not tolerate the insertion of the I-Gel, an extra dose of fentanyl up to a maximum of 0.5 mcg / kg in total was administered. However, if the insertion attempt was still not tolerated, or if the capnography curve was not obtained and there was an audible leak, the technique was considered to be unsuccessful, and another SGA was then placed in the airway. If this change was not tolerated, endotracheal intubation was initiated by applying neuromuscular blocker and these were recorded.

USG examination of the neck was performed by the second anesthesiologist using an 8-18 MHz linear probe Esaote Imaging was done in three planes (Transverse plane between hyoid bone and thyroid bone, Transverse plane of the lateral suprasternal notch and Parasagittal plane of pharynx and larynx) the USG score was assigned to the deployment view using a modification of the criteria proposed.

The fiberoptic bronchoscope was passed through I-Gel until the glottis image was obtained.Optimal placement was defined as the end of the I-Gel behind the arytenoids, with a visible epiglottis, with or without folding to the airway, and the vocal cords are visible when the FOB is advanced under the epiglottis.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing elective pediatric surgery
* American Society of Anesthesiologists (ASA) status I-II
* Placed I-Gel for airway

Exclusion Criteria:

* Patients with head and neck anatomical malformation and airway congenital defects

Ages: 1 Month to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The pediatric patients who were scheduled to undergo surgery under general anesthesia placed I-Gel for airway were enrolled in the study.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2020-12-15 (Estimated); Primary Completion 2021-01-30 (Estimated); Study Completion 2021-02-15 (Estimated)

PRIMARY OUTCOMES:
the incidence of for I-Gel malposition between USG and FOB | 1 months
  to compare the incidence of for I-Gel malposition between USG and FOB.

SECONDARY OUTCOMES:
the correlation between I-Gel's USG and FOB | 1 months
  to find the correlation between I-Gel's USG and FOB-detected malposition and to determine the diagnostic performance of the USG.

CONTACTS AND LOCATIONS:
Overall Officials: Faruk Cicekci, Principal Investigator — Selcuk University, School of Medicine, Department of Anesthesiology and Intensive Care
Locations (1):
- Selcuk University, School of Medicine, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No